CLINICAL TRIAL: NCT04609501
Title: Delivery During Covid-19 Pandemic: Implications for Obstetrics, Maternal Psychopathology, and Mother-Infant Relationship in the Shadow of a Socioeconomic Crisis
Brief Title: Delivery During Covid-19 Pandemic: Implications for Obstetrics, Maternal Psychopathology, and Mother-Infant Relationship
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: 0082-20-HYMC
Record Dates: First submitted 2020-10-22; First posted 2020-10-30 (Actual); Last update posted 2022-06-23 (Actual); Status verified 2022-06

CONDITIONS: Delivery; Trauma; Covid19
MeSH Terms: conditions — Wounds and Injuries; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Coronavirus 2019 (COVID-19) pandemic has brought about unprecedented social, economic and mental-health challenges, especially for vulnerable populations such as pregnant and post-partum females. In this study, we aimed to evaluate the relations between the fear of COVID-19 and postnatal depression symptoms.

DETAILED DESCRIPTION:
This is a multicenter prospective cohort study of childbearing women during COVID-19. Participants completed a comprehensive online questionnaire including demographic, socioeconomic, obstetric, and postnatal mental-health questionnaires. Data were verified with each center's perinatal database and information regarding physiological stress during pregnancy/birth was also collected. Fear of COVID-19 was evaluated using the validated Fear of COVID-19 Scale and postnatal depression was evaluated using the EPDS. Pre-existing maternal disability was defined as prior physiological or psychological chronic health condition.

ELIGIBILITY:
Inclusion Criteria:

* women who delivered during the Covid-19 pandemic at the site, since 01-March-2020

Exclusion Criteria:

* women age 18 and below
* Gestational age under 34 weeks
* Intra Uterine Fetal Demise
* Ante-partum Fetal Demise
* Maternal post partum death

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Women after delivery
Study Population: women who delivered during the Covid-19 pandemic
Sampling Method: Non-Probability Sample
Enrollment: 440 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Evaluation of COVID-19 during pregnancy | 1 year after delivery
  Fear of COVID-19 was evaluated using the validated Fear of COVID-19 Scale
The relations between fear of COVID-19 and postnatal depression symptoms. | 1 year after delivery
  Postnatal depression was evaluated using the EPDS.

CONTACTS AND LOCATIONS:
Overall Officials: Rinat Gabbay-Benziv, MD, Principal Investigator — Hillel Yaffe Medical Center
Locations (1):
- Department of Obstetrics and Gynecology, Hillel-Yaffe Medical Center, Hadera, Israel